CLINICAL TRIAL: NCT06441110
Title: Multicentre Clinical Trial of the Efficacy and Safety of Tislelizumab in Combination With BCG Bladder Instillation in the Prevention of Postoperative Recurrence in Intermediate and High-risk Non-muscle Invasive Bladder Cancer
Brief Title: Multicenter Clinical Trial on the Effectiveness and Safety of Instillation of BCG and Alternative BCG Protocols for Intermediate and High-risk Non-muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023XHYG0045-02
Record Dates: First submitted 2024-05-14; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-04

CONDITIONS: Urinary Bladder Neoplasms; BCG Vaccine; Immunotherapy, Active; Multicenter Study; Treatment Outcome; Neoplasm Recurrence, Local
MeSH Terms: conditions — Urinary Bladder Neoplasms; Motor Activity; Neoplasm Recurrence, Local | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postoperative Instillation Therapy Group (Experimental): Tislelizumab in Combination with Bacillus Calmette-Guérin for the Treatment of Intermediate and High-Risk NMIBC Group
  Interventions: Drug: Tislelizumab in Combination with Bacillus Calmette-Guérin

INTERVENTIONS:
Drug: Tislelizumab in Combination with Bacillus Calmette-Guérin — Postoperative immediate instillation of epirubicin (50mg) is administered. Postoperatively, 200mg of tislelizumab injection is given intravenously every 3 weeks, with each 21-day period constituting one cycle. The medication is administered on day 1 of each cycle, continuing for one year. Eligible patients for the single-arm group (N = 76) begin BCG instillation after 2 weeks, with a dosage of 120mg per instillation, totaling 19 instillations: this starts with a 6-week induction phase of weekly BCG instillations, followed by BCG instillations every 2 weeks for three consecutive times; thereafter, maintenance instillation therapy commences, involving monthly BCG instillations for a total of ten times.

SUMMARY:
Previous studies have reported the efficacy of Bacillus Calmette-Guérin (BCG) combined with other drugs for the treatment of bladder cancer. However, research on the combination of tislelizumab and BCG for bladder cancer treatment has largely been retrospective. Currently, ongoing clinical trials have not discussed the effectiveness of PD-1/PD-L1 inhibitors combined with BCG instillation in reducing postoperative recurrence in intermediate-risk NMIBC. Therefore, this study aims to explore the clinical efficacy and safety of tislelizumab combined with BCG in the treatment of intermediate and high-risk NMIBC. For this purpose, investigators have established strict screening criteria to include eligible patients in the study and have recruited suitable patients from multiple medical centers.Investigators have also developed a meticulous implementation process and follow-up considerations, hoping to better verify the clinical efficacy and safety of the combined use of these two drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the trial with signed informed consent;
2. Patients aged ≥18 and ≤75 years, regardless of gender, with an expected survival of ≥2 years;
3. Histologically confirmed non-muscle-invasive bladder urothelial carcinoma with positive PD-L1 expression. According to the 2014 guidelines of the Chinese Urological Association (CUA), patients are assessed as having a medium to high risk of recurrence or progression. (For patients considering a second transurethral resection, they may be included in the study after completing the procedure and if pathology confirms medium to high risk non-muscle-invasive bladder urothelial carcinoma);
4. Performance status score (Eastern Cooperative Oncology Group, ECOG) of 0-2;
5. Completion of screening-related examinations (complete blood count, coagulation function, liver and kidney function, infectious disease screening, 12-lead ECG, urinary system ultrasound, pelvic MR, and tissue pathology examination), without surgical contraindications.

Exclusion Criteria:

1. Any of the following conditions:

   Immune deficiency or impairment (such as AIDS patients), current use of immunosuppressive drugs or radiation therapy that may cause systemic BCG disease reaction; allergy to BCG components; patients with fever and acute infectious diseases, including active tuberculosis or those undergoing anti-tuberculosis treatment; those with severe chronic cardiovascular or cerebrovascular diseases or chronic kidney disease;
2. Concurrent urogenital system tumors or tumors in other organs;
3. Muscle-invasive bladder urothelial carcinoma (stage T2 and above) patients;
4. Patients who have received chemotherapy, radiotherapy, or immunotherapy within the past 4 weeks (except immediate postoperative bladder instillation chemotherapy);
5. Pregnant or lactating women, women of childbearing age not using effective contraception, or those planning to conceive during the trial period (including male participant partners);
6. Known or suspected intraoperative bladder perforation;
7. Presence of gross hematuria prior to enrollment, suspected unhealed surgical wounds or damaged urinary mucosa;
8. Severe urethral stricture preventing cystoscopy, history of bladder contracture, or functional bladder volume less than 100mL;
9. Accompanying cystitis, or those who have received other bladder instillation medications and have severe bladder irritation signs expected to affect the assessment of this study;
10. Patients with various mental disorders, severe coagulation function, liver and kidney function, hematopoietic function disorders, etc., that cannot tolerate surgical treatment;
11. Participation in other drug clinical trials within 3 months before enrollment;
12. Known or suspected opioid or alcohol dependence;
13. Any condition that the researcher believes may increase the risk to the participant or interfere with the execution of the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2035-06-01 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival(RFS) | From date of postoperative cystoscopic examination to the first documented recurrence of bladder tumor,assessed up to 60 months.
  The time from postoperative cystoscopic examination to the first documented recurrence of bladder tumor.

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | From date of postoperative cystoscopic and pathological examinations to the first progression of bladder tumor, assessed up to 60 months.
  The time recorded from postoperative cystoscopic and pathological examinations to the first progression of bladder tumor, defined in this trial as the occurrence of muscle-invasive growth in NMIBC (Non-Muscle Invasive Bladder Cancer) patients.
Overall survival | From date of post-surgery to the time of death due to any cause,assessed up to 60 months
  The duration from post-surgery to the time of death due to any cause. For participants who are lost to follow-up prior to death, the time of their last follow-up is typically considered as the time of death for calculation purposes.
Adverse event（AS) | From date of post-surgery to the time of death due to any cause,assessed up to 60 months.
  An adverse event (AE) is defined according to the toxicity grading standards set by the National Cancer Institute of the United States. This includes a spectrum of adverse reactions associated with antineoplastic therapy. Specific grading of adverse reactions refers to the Common Terminology Criteria for Adverse Events (CTCAE Version 5.0) developed by the National Cancer Institute (NCI).

CONTACTS AND LOCATIONS:
Overall Officials: Zhenlin Chen, Principal Investigator — Department of Urology, Fujian Union Hospital, Fujian Medical University
Locations (1):
- Department of Urology, Fujian Union Hospital, Fujian Medical University, Fuzhou, Fujian, China